CLINICAL TRIAL: NCT06661473
Title: An Interventional Study to Explore the Occurrence of Surgical Site Complications in High-risk Patients After Revision of Total Hip or Knee Joint Arthroplasty Receiving Closed Incision Negative Pressure Wound Therapy.
Brief Title: Interventional Study Exploring the Occurrence of Surgical Site Infections.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Asolo SSC
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty; Total Hip Arthroplasty Revision; Total Knee Arthroplasty Revision
Keywords: high risk TKA revision; high risk THA revision; NPWT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Avance Solo ciNPT (Other)
  Interventions: Device: Avance Solo Negative Pressure Wound Therapy

INTERVENTIONS:
Device: Avance Solo Negative Pressure Wound Therapy — Avance Solo NPWT 7-14 days after high-risk revision TKA or THA.

SUMMARY:
Interventional study exploring surgical site complication occurrences in high-risk revision patients undergoing TKA or THA using NPWT.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Patient ≥ 18 years
3. Elective unilateral revision THA or TKA.
4. High risk patients for surgical wound complications as deemed by investigators
5. Primary closure technique by suture or staples
6. Linear or curvilinear incisions ≤ 25 cm in length
7. The patient able to understand the study and is willing to consent to the clinical investigation
8. Patients able to understand how to operate with the negative pressure system at home

Exclusion Criteria:

1. The need for emergency surgery
2. Multiple Incision Approach at the time of surgery (alternative approach from primary surgery using 1 incision is permitted)
3. Patients requiring bilateral revision total hip or knee arthroplasty surgery
4. Active infections of the offending joint.
5. History of multiple infections in the offending joint
6. Patients with known allergies to product components (silicone adhesives and polyurethane films (direct contact with wound), acrylic adhesives (direct contact with skin), polyethylene fabrics and superabsorbent powders (polyacrylates) (within the dressing)
7. Subjects with contraindications (as per the Avance Solo Instructions for use)
8. Pregnant, breastfeeding females, or females of childbearing potential not willing to use contraception for the duration of the investigation
9. Patients with presence of remote skin infection or active systemic infection at the time of revision surgery.
10. Patient with incisions > 25cm in length or type of incisions that cannot be sufficiently covered by Avance Solo Border dressing (i.e., the wound pad does not overlap the edges of the incision by at least 1.5 cm as per the IFU)
11. Use of surgical glue as part of incisional closure method
12. Patients who in the opinion of the investigator may not complete or comply with follow up treatment for any reason
13. Patients participating in ongoing clinical investigations, or during the past 30 days, that may impact the outcome of this investigation based on the judgement of the investigator.
14. Any clinically significant condition that, in the investigator's opinion, would significantly impair the subject's ability to comply with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infections | 90 days from revision surgery

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - MedStar Health, Washington D.C., District of Columbia
  - Ortho Indy, Indianapolis, Indiana
  - Life Bridge Health- Sinai Hospital, Baltimore, Maryland
  - Twin Cities Orthopedics, Minneapolis, Minnesota
  - St. Louis University, St Louis, Missouri
  - Northwell, Garden City, New York
  - Bon Secours Mercy Health, Youngstown, Ohio
  - Spokane Joint Replacement Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No